CLINICAL TRIAL: NCT03726489
Title: A Pragmatic Trial of Home Versus Office Based Narrow Band Ultraviolet B Phototherapy for the Treatment of Psoriasis
Brief Title: Light Treatment Effectiveness (LITE) Study
Acronym: LITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Utah (Other); National Psoriasis Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 831323; PCS-1608-35830 (Other Grant/Funding Number: Patient-Centered Outcomes Research Insitute)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis; Psoriatic Plaque
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Pragmatic, randomized, active comparator effectiveness study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Office Based Phototherapy (Other): Patients randomized to this arm will receive narrow band phototherapy in a clinical setting via narrow band phototherapy clinic units.
  Interventions: Device: narrow band phototherapy clinic units
- Home Based Phototherapy (Active Comparator): Patients randomized to this arm will receive narrow band phototherapy in a home setting via Daavlin 7 series 3 panel narrow band phototherapy home units.
  Interventions: Device: Daavlin 7 series 3 panel narrow band phototherapy home units

INTERVENTIONS:
Device: Daavlin 7 series 3 panel narrow band phototherapy home units — Daavlin 7 series 3 panel narrow band phototherapy home units (with 8-12 bulbs and a smaller, flat surface with door, measuring 21" wide, 74.5" tall, and 23.5"). This unit is a class II device with a FDA 510K indication for psoriasis, vitiligo and atopic dermatitis/eczema. The unit will have a dosimetry controller, a UV sensor built in that measures the intensity of the light. This sensor will adjust the treatment time to compensate for any variation in output due to aging of the lamps or other factors
  Arms: Home Based Phototherapy
Device: narrow band phototherapy clinic units — Office based narrow band phototherapy unit (units typically have at least 24 bulbs in a surround structure
  Arms: Office Based Phototherapy

SUMMARY:
To compare the effectiveness, safety (tolerability), and duration of treatment response at 12 weeks of home versus office-based narrowband ultraviolet B phototherapy for the treatment of psoriasis

DETAILED DESCRIPTION:
The primary objective of this study is to compare the effectiveness, safety (tolerability), and duration of treatment response at 12 weeks of home versus office-based narrowband ultraviolet B phototherapy for the treatment of psoriasis. Physician Global Assessment (PGA) and Dermatology Life Quality Index (DLQI) will be used to assess effectiveness, safety (tolerability), and duration of treatment response. This is a three year pragmatic, randomized, active comparator effectiveness study.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent (age 18+) or parental permission and assent (ages 12-17)
2. Age 12 or older
3. Plaque or guttate psoriasis predominantly located on trunk and/or extremities, with a physician global assessment average of >1.0, and considered a candidate for phototherapy
4. Patient is deemed willing and able to comply with either in-office or in-home phototherapy:

   1. In office: Able to travel about 3 times per week for 12 weeks from home, work and/or school during business hours of local site
   2. In home: Has space to accommodate home phototherapy unit and patient (or if 12-17, parent), willing and able to follow home phototherapy instructions
5. New or established patient in the practice

Exclusion Criteria:

1. Patients who are judged unable or unwilling to comply with either in office or in home phototherapy due to time, work, school, or other financial constraints
2. Patients judged unable to follow home phototherapy protocol due to failure to demonstrate understanding of the following:

   1. How to operate the phototherapy device
   2. How to follow the dosing protocol
   3. Requirement to wear protective eyewear and genital protection equipment
3. Patients with known history of lack of efficacy to phototherapy or treated with phototherapy 14 days prior to baseline visit
4. Psoriasis predominantly located on scalp, body folds, genitals, palms and/or soles or with a physician global assessment average of ≤ 1.0
5. Patients deemed unsafe to be treated with phototherapy:

   1. History of photosensitivity or autoimmune disease such as lupus or dermatomyositis which can be aggravated by ultraviolet radiation
   2. History of arsenic intake
   3. Unable to tolerate standing for required duration of treatment due to age or physical function
   4. History of melanoma or multiple non-melanoma skin cancers that in the opinion of the principal investigator contraindicates treatment with phototherapy
6. Clinical site deems the participant is ineligible for reason other than eligibility or screening criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M. Gelfand, MD,MSCE, Principal Investigator — University of Pennsylvania
Locations (38):
- United States (38):
  - Total Skin & Beauty Dermatology Center, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - University of Southern California, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Dawes Fretzin Clinical Research, Indianapolis, Indiana
  - MD Claiborne and Associates, LLC, New Orleans, Louisiana
  - MaineHealth/Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - DermAssociates LLC, Silver Spring, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dermatology Specialist of Brighton, Brighton, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Heymann, Manders, Green, and Sommer, LLC, Marlton, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - HHC Kings County Hospital, Brooklyn, New York
  - SUNY Downstate Health Sciences University, Brooklyn, New York
  - Buffalo Medical Group, Buffalo, New York
  - Infinity Dermatology NYC, Queens, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Pennsyvlania Centre For Dermatology, Exton, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - West Houston Dermatology, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont & State Agriculture College, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Gelfand JM, Armstrong AW, Lim HW, Feldman SR, Johnson SM, Claiborne WCC, Kalb RE, Jakus J, Mangold AR, Flowers RH, Bhutani T, Durkin JR, Bagel J, Fretzin S, Sheehan MP, Krell J, Reeder M, Kaffenberger J, Kartono F, Takeshita J, Bridges AM, Fielding E, Nehal US, Schaecher KL, Howard LM, Eakin GS, Baez S, Bishop BE, Fitzsimmons RC Jr, Papadopoulos M, Song WB, Linn KA, Hubbard RA, Shin DB, Callis Duffin K. Home- vs Office-Based Narrowband UV-B Phototherapy for Patients With Psoriasis: The LITE Randomized Clinical Trial. JAMA Dermatol. 2024 Dec 1;160(12):1320-1328. doi: 10.1001/jamadermatol.2024.3897. PMID 39319513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Started | 390 | 393
Received Phototherapy (Subjects who initiated phototherapy) | 232 | 309
DLQI Assessed (Includes subjects who completed DLQI before or within assessment window.) | 252 | 308
PGA Assessed | 217 | 255
Completed (Includes subjects who withdrew prior to Week 12, who are included in the analysis as non-responders) | 390 | 393
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Office Based Phototherapy | Home Based Phototherapy | Total
Number analyzed (Participants) | 390 | 393 | 783
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.1) | 48.2 (15.9) | 48.0 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 186 | 376
  Male | 200 | 207 | 407
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 48 | 102
  Not Hispanic or Latino | 328 | 334 | 662
  Unknown or Not Reported | 8 | 11 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 292 | 296 | 588
  Race: Black | 34 | 39 | 73
  Race: Asian | 31 | 25 | 56
  Race: Other | 33 | 33 | 66
Skin Phototype [Count of Participants; unit: Participants] — Stratification variable based on Fitzpatrick skin phototype. The Fitzpatrick scale is a numerical classification schema for human skin color. It was developed as a way to estimate the response of different types of skin to ultraviolet (UV) light. The scale ranges from Type I (always burns, never tans, pale) to Type VI (never burns, i.e. deeply pigmented dark brown to darkest brown).
  Participants
    I/II | 169 | 181 | 350
    III/IV | 180 | 170 | 350
    V/VI | 41 | 42 | 83
Estimated time traveling to/from phototherapy treatment [Mean (Standard Deviation); unit: minutes] — Population: Missing data due to survey non-response
  minutes
    number analyzed (Participants) | 328 | 324 | 652
    (all) | 59.1 (50.6) | 58.0 (42.3) | 58.5 (46.6)
Estimated time traveling to/from dermatologist office [Mean (Standard Deviation); unit: minutes] — Population: Missing data due to survey non-response
  minutes
    number analyzed (Participants) | 328 | 324 | 652
    (all) | 58.2 (47.0) | 61.3 (49.1) | 59.8 (48.1)
Miles from dermatologist office [Mean (Standard Deviation); unit: miles] — Population: Missing data due to non-response
  miles
    number analyzed (Participants) | 328 | 324 | 652
    (all) | 30.68 (35.21) | 32.26 (26.19) | 31.48 (36.98)
Co-pay for dermatologist [Mean (Standard Deviation); unit: USD] — Population: Missing data due to survey non-response
  USD
    number analyzed (Participants) | 385 | 388 | 773
    (all) | 22.3 (31.9) | 21.0 (30.3) | 21.6 (31.1)
Co-pay for phototherapy treatment [Mean (Standard Deviation); unit: USD] — Population: Missing data due to survey non-response
  USD
    number analyzed (Participants) | 385 | 388 | 773
    (all) | 17.5 (30.5) | 17.5 (30.4) | 17.5 (30.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (7.6) | 29.3 (6.8) | 29.6 (7.2)
Medical history [Count of Participants; unit: Participants]
  Psoriatic arthritis present | 65 | 68 | 133
  History of internal malignancy | 27 | 21 | 48
  History of skin cancer | 4 | 7 | 11
  History of cardiovascular disease | 25 | 27 | 52
  History of diabetes | 43 | 40 | 83
  History of hypertension | 91 | 96 | 187
  History of hyperlipidemia | 56 | 57 | 113
  History of arthritis | 19 | 25 | 44
  History of mood disorder | 37 | 38 | 75
  History of anxiety | 32 | 30 | 62
  History of mood disorder/anxiety | 58 | 54 | 112
  Pregnant | 0 | 1 | 1
  History of cardiometabolic disease | 221 | 233 | 454
Baseline DLQI [Mean (Standard Deviation); unit: units on a scale (0-30)] — Dermatology Life Quality Index (DLQI) consists of 10 questions that ask about symptoms, feelings, daily activities, leisure, work, school, personal relationships, and treatment. Each question is scored from 0 to 3, with "not at all" being 0, "a little" being 1, "quite a lot" being 2, and "very much" being 3. The total score ranges from 0 to 30, with higher scores indicating a greater impairment of quality of life. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease. Population: Missing data due to survey non-response
  units on a scale (0-30)
    number analyzed (Participants) | 349 | 344 | 693
    (all) | 12.3 (7.2) | 12.1 (7.3) | 12.2 (7.2)
Baseline PGA [Mean (Standard Deviation); unit: units on a scale] — The Physician's Global Assessment is an average assessment of all psoriatic lesions based on three components (erythema, scale, and induration) ranging from 0 (no evidence of disease) to 5 (maximal disease). All components are individually assessed and averaged for the PGA value.
  units on a scale | 2.7 (0.8) | 2.7 (0.8) | 2.7 (0.8)
BSA [Mean (Standard Deviation); unit: percentage] — Body surface area (%) affected
  percentage | 12.4 (15.3) | 12.6 (16.1) | 12.5 (15.7)
Age at psoriasis diagnosis [Mean (Standard Deviation); unit: years] | 32.4 (17.5) | 32.0 (18.8) | 32.2 (18.2)
Psoriasis duration [Mean (Standard Deviation); unit: years] | 15.4 (14.6) | 16.2 (15.0) | 15.8 (14.8)
Treatment history [Count of Participants; unit: Participants]
  Biologics | 84 | 83 | 167
  Non-biological systemic therapy | 110 | 121 | 231
  Biologics or non-biological systemic therapy | 155 | 157 | 312
  Phototherapy | 165 | 172 | 337
Current treatment [Count of Participants; unit: Participants]
  Biologics | 30 | 25 | 55
  Non-biological systemic therapy | 24 | 21 | 45
  Biologics or non-biological systemic therapy | 49 | 44 | 93

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Assessment (PGA) Score of Clear/Almost Clear
Description: Measure of clinical treatment response, with PGA score of 0/1 (clear/almost clear). PGA score range from 0 (clear) to 5 (worst disease state).
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: The outcome measures were analyzed by skin phototype strata in addition to total subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 390 | 393
Participants
  All phototypes | 100 | 129
  Phototype I/II: number analyzed (Participants) | 169 | 181
  Phototype I/II | 47 | 58
  Phototype III/IV: number analyzed (Participants) | 180 | 170
  Phototype III/IV | 47 | 57
  Phototype V/VI: number analyzed (Participants) | 41 | 42
  Phototype V/VI | 6 | 14
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis including all skin phototypes; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; Test statistic is based on risk difference and standard error calculated using marginal standardization from adjusted logistic regression estimates; Risk Difference (RD) = 7.2, 95% CI 2-sided [0.8 to 13.5]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 4.2, 95% CI 2-sided [-5.4 to 13.8]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 7.4, 95% CI 2-sided [-2.2 to 17.0]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%. The sample size for this subgroup did not meet our a priori sample size required for 80% power; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 18.7, 95% CI 2-sided [0.8 to 36.6]
Statistical Analysis 5: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for heterogeneity of treatment effects (HTE) including all skin phototypes; Test type: Other — HTE was assessed using an omnibus Wald test of all interaction regression parameters in order to minimize multiple testing and consequent alpha inflation; p = 0.347, Regression, Logistic — HTE was assessed using an omnibus Wald test of all interaction regression parameters in order to minimize multiple testing and consequent alpha inflation; We fit models for each of the two primary outcomes with skin type, treatment arm, and their interaction as predictors

2. Primary Outcome: Impact of Dermatological Disease on Quality of Life (DLQI ≤5)
Description: Dermatology Life Quality Index (DLQI) score of ≤5 which corresponds to no to small impact of dermatologic disease on quality of life. DLQI is a 10 item survey that asks patients questions about their health related quality of life on a 0-3 scale. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: The outcome measures were analyzed by skin phototype strata in addition to total subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 390 | 393
Participants
  All phototypes | 131 | 206
  Phototype I/II: number analyzed (Participants) | 169 | 181
  Phototype I/II | 65 | 108
  Phototype III/IV: number analyzed (Participants) | 180 | 170
  Phototype III/IV | 56 | 81
  Phototype V/VI: number analyzed (Participants) | 41 | 42
  Phototype V/VI | 10 | 17
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis including all skin phototypes; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 18.6, 95% CI 2-sided [11.8 to 25.3]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 21.2, 95% CI 2-sided [11.0 to 31.5]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 16.5, 95% CI 2-sided [6.4 to 26.6]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 4]; p = 0.001, Marginal standardization — P-value was not adjusted for multiple comparisons. All p-values below 0.001 are reported as <0.001; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 16.1, 95% CI 2-sided [-3.7 to 35.9]
Statistical Analysis 5: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for heterogeneity of treatment effects (HTE) including all skin phototypes; Test type: Other; p = 0.873, Regression, Logistic — [p-value comment as in outcome 1, analysis 5]; We fit models for each of the two primary outcomes with skin type, treatment arm, and their interaction as predictors

3. Secondary Outcome: Total Number of Phototherapy Treatments Received
Description: patient or site reported phototherapy dosing
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: The outcome measures were analyzed by skin phototype strata in addition to total subjects. Participants with missing data were excluded from the overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: treatments
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 232 | 309
treatments
  All phototypes | 17.95 (8.83) | 26.82 (10.63)
  Phototype I/II: number analyzed (Participants) | 105 | 153
  Phototype I/II | 18.86 (8.99) | 28.24 (9.57)
  Phototype III/IV: number analyzed (Participants) | 103 | 129
  Phototype III/IV | 17.72 (8.49) | 26.20 (11.40)
  Phototype V/VI: number analyzed (Participants) | 24 | 27
  Phototype V/VI | 14.96 (9.15) | 21.78 (11.07)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [7.1 to 10.4]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 9.38, 95% CI 2-sided [7.05 to 11.71]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 8.48, 95% CI 2-sided [5.82 to 11.14]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.0213, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 6.82, 95% CI 2-sided [1.06 to 12.58]

4. Secondary Outcome: Cumulative Dose of Phototherapy Received
Description: Cumulative dose of photherapy is the sum of all individual doses from randomization to week 12 visit.
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: J/cm^2
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 232 | 309
J/cm^2
  All phototypes | 17.27 (16.09) | 31.43 (29.55)
  Phototype I/II: number analyzed (Participants) | 105 | 153
  Phototype I/II | 15.04 (13.19) | 26.51 (20.94)
  Phototype III/IV: number analyzed (Participants) | 103 | 129
  Phototype III/IV | 18.93 (16.79) | 32.80 (27.64)
  Phototype V/VI: number analyzed (Participants) | 24 | 27
  Phototype V/VI | 19.90 (22.86) | 52.73 (58.29)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = 14.6, 95% CI 2-sided [10.4 to 18.7]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 11.47, 95% CI 2-sided [6.93 to 16.01]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p < 0.0001, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 13.87, 95% CI 2-sided [7.77 to 19.98]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.0127, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 32.84, 95% CI 2-sided [7.32 to 58.35]

5. Secondary Outcome: Concomitant Topical Psoriasis Treatment
Description: Patient reported topical psoriasis treatment - number of days per week the patient takes topical medication
Time Frame: week 12 and week 24 after randomization
Population: The outcome measures were analyzed by skin phototype strata in addition to total subjects
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 269 | 325
days per week
  All phototypes | 3.92 (2.91) | 3.06 (2.80)
  Phototype I/II: number analyzed (Participants) | 110 | 159
  Phototype I/II | 3.61 (2.91) | 2.77 (2.67)
  Phototype III/IV: number analyzed (Participants) | 128 | 136
  Phototype III/IV | 4.02 (2.85) | 3.13 (2.88)
  Phototype V/VI: number analyzed (Participants) | 31 | 30
  Phototype V/VI | 4.65 (3.06) | 4.23 (2.88)
  All phototypes (week 24): number analyzed (Participants) | 160 | 215
  All phototypes (week 24) | 3.59 (2.74) | 3.34 (2.81)
  Phototype I/II (week 24): number analyzed (Participants) | 70 | 112
  Phototype I/II (week 24) | 3.46 (2.67) | 3.34 (2.71)
  Phototype III/IV (week 24): number analyzed (Participants) | 76 | 85
  Phototype III/IV (week 24) | 3.74 (2.78) | 3.21 (2.88)
  Phototype V/VI (week 24): number analyzed (Participants) | 14 | 18
  Phototype V/VI (week 24) | 3.50 (3.01) | 3.94 (3.21)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.001, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.27 to -0.35]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.0158, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.51 to -0.16]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.0130, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.58 to -0.19]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.5910, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-1.94 to 1.11]
Statistical Analysis 5: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes at Week 24; Test type: Superiority; p = 0.395, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = .25, 95% CI 2-sided [-0.33 to 0.82]
Statistical Analysis 6: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II at Week 24; Test type: Superiority; p = 0.774, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.69 to 0.93]
Statistical Analysis 7: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV at Week 24; Test type: Superiority; p = 0.242, Regression, Linear — P-value was not adjusted for multiple comparisons; Median Difference (Final Values) = 0.53, 95% CI 2-sided [-0.36 to 1.41]
Statistical Analysis 8: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI at Week 24; Test type: Superiority; p = 0.692, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-2.72 to 1.83]

6. Secondary Outcome: Changes in Initiation or Discontinuation of Oral or Biologic Psoriasis Treatments
Time Frame: week 12 and week 24 after randomization
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 317 | 339
Participants
  All phototypes - Initiation: number analyzed (Participants) | 280 | 308
  All phototypes - Initiation | 16 | 9
  Phototype I/II - Initiation: number analyzed (Participants) | 114 | 145
  Phototype I/II - Initiation | 4 | 2
  Phototype III/IV - Initiation: number analyzed (Participants) | 133 | 134
  Phototype III/IV - Initiation | 10 | 6
  Phototype V/VI - Initiation: number analyzed (Participants) | 33 | 29
  Phototype V/VI - Initiation | 2 | 1
  All phototypes - Discontinuation: number analyzed (Participants) | 280 | 308
  All phototypes - Discontinuation | 8 | 9
  Phototype I/II - Discontinuation: number analyzed (Participants) | 114 | 145
  Phototype I/II - Discontinuation | 2 | 3
  Phototype III/IV - Discontinuation: number analyzed (Participants) | 133 | 134
  Phototype III/IV - Discontinuation | 5 | 6
  Phototype V/VI - Discontinuation: number analyzed (Participants) | 33 | 29
  Phototype V/VI - Discontinuation | 1 | 0
  All phototypes - Initiation (Week 24) | 31 | 28
  Phototype I/II - Initiation (Week 24): number analyzed (Participants) | 136 | 162
  Phototype I/II - Initiation (Week 24) | 9 | 10
  Phototype III/IV - Initiation (Week 24): number analyzed (Participants) | 145 | 145
  Phototype III/IV - Initiation (Week 24) | 17 | 14
  Phototype V/VI - Initiation (Week 24): number analyzed (Participants) | 36 | 32
  Phototype V/VI - Initiation (Week 24) | 5 | 4
  All phototypes - Discontinuation (Week 24) | 8 | 9
  Phototype I/II - Discontinuation (Week 24): number analyzed (Participants) | 136 | 162
  Phototype I/II - Discontinuation (Week 24) | 2 | 3
  Phototype III/IV - Discontinuation (Week 24): number analyzed (Participants) | 145 | 145
  Phototype III/IV - Discontinuation (Week 24) | 5 | 6
  Phototype V/VI - Discontinuation (Week 24): number analyzed (Participants) | 36 | 32
  Phototype V/VI - Discontinuation (Week 24) | 1 | 0
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes - Initiation; Test type: Superiority; p = 0.1209, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -2.59, 95% CI 2-sided [-5.86 to 0.68]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II - Initiation; Test type: Superiority; p = 0.2581, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -2.13, 95% CI 2-sided [-6.0 to 1.75]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV - Initiation; Test type: Superiority; p = 0.2952, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -3.04, 95% CI 2-sided [-8.73 to 2.65]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI - Initiation; Test type: Superiority; p = 0.6324, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -2.61, 95% CI 2-sided [-13.12 to 7.89]
Statistical Analysis 5: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes - Discontinuation; Test type: Superiority; p = 0.9163, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.15, 95% CI 2-sided [-2.56 to 2.85]
Statistical Analysis 6: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II - Discontinuation; Test type: Superiority; p = 0.8551, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.31, 95% CI 2-sided [-3.03 to 3.66]
Statistical Analysis 7: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV - Discontinuation; Test type: Superiority; p = 0.7678, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.72, 95% CI 2-sided [-4.05 to 5.48]
Statistical Analysis 8: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI - Discontinuation; Test type: Superiority; p = 0.3446, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -3.03, 95% CI 2-sided [-8.88 to 2.82]
Statistical Analysis 9: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes - Initiation at Week 24; Test type: Superiority; p = 0.5716, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -1.26, 95% CI 2-sided [-5.64 to 3.11]
Statistical Analysis 10: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II - Initiation at Week 24; Test type: Superiority; p = 0.8756, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -0.44, 95% CI 2-sided [-6.03 to 5.14]
Statistical Analysis 11: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV - Initiation at Week 24; Test type: Superiority; p = 0.5686, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -2.07, 95% CI 2-sided [-9.18 to 5.04]
Statistical Analysis 12: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI - Initiation at Week 24; Test type: Superiority; p = 0.8660, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -1.39, 95% CI 2-sided [-17.5 to 14.7]
Statistical Analysis 13: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes - Discontinuation at Week 24; Test type: Superiority; p = 0.8779, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.19, 95% CI 2-sided [-2.24 to 2.62]
Statistical Analysis 14: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II - Discontinuation at Week 24; Test type: Superiority; p = 0.7985, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.38, 95% CI 2-sided [-2.52 to 3.28]
Statistical Analysis 15: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV - Discontinuation at Week 24; Test type: Superiority; p = 0.7585, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 0.69, 95% CI 2-sided [-3.71 to 5.09]
Statistical Analysis 16: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI - Discontinuation at Week 24; Test type: Superiority; p = 0.3422, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -2.78, 95% CI 2-sided [-8.15 to 2.59]

7. Secondary Outcome: Patient-reported Time Spent on Phototherapy Per Treatment
Description: patient reported survey
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 190 | 242
minutes
  All phototypes | 21.8 (18.2) | 18.5 (20.9)
  Phototype I/II: number analyzed (Participants) | 79 | 112
  Phototype I/II | 21.58 (20.45) | 16.32 (14.59)
  Phototype III/IV: number analyzed (Participants) | 93 | 109
  Phototype III/IV | 22.03 (16.77) | 18.11 (21.14)
  Phototype V/VI: number analyzed (Participants) | 18 | 21
  Phototype V/VI | 22.06 (15.09) | 32.48 (38.13)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.094, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = -3.20, 95% CI 2-sided [-6.95 to 0.55]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.0393, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -5.26, 95% CI 2-sided [-10.26 to -0.26]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.1505, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -3.92, 95% CI 2-sided [-9.28 to 1.44]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.2840, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 10.42, 95% CI 2-sided [-9.0 to 29.84]

8. Secondary Outcome: Patient Reported Costs Associated With Travel for Phototherapy Treatments
Description: patient reported survey for Office patients only
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Office Based Phototherapy
Number analyzed (Participants) | 190
USD
  All phototypes | 19.9 (61.6)
  Phototype I/II: number analyzed (Participants) | 79
  Phototype I/II | 18.06 (57.04)
  Phototype III/IV: number analyzed (Participants) | 93
  Phototype III/IV | 23.46 (70.71)
  Phototype V/VI: number analyzed (Participants) | 18
  Phototype V/VI | 9.22 (5.66)
Statistical Analysis 1: Comparison: Office Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Other; P-value is not applicable; Mean = 19.87, Standard Deviation 61.6
Statistical Analysis 2: Comparison: Office Based Phototherapy; Analysis for Phototypes I/II; Test type: Other; P-value is not applicable; Mean = 18.06, Standard Deviation 57.04
Statistical Analysis 3: Comparison: Office Based Phototherapy; Analysis for Phototypes III/IV; Test type: Other; P-value is not applicable; Mean = 23.46, Standard Deviation 70.71
Statistical Analysis 4: Comparison: Office Based Phototherapy; Analysis for Phototypes V/VI; Test type: Other; P-value is not applicable; Mean = 9.22, Standard Deviation 5.66

9. Secondary Outcome: Patient Reported Time Associated With Travel for Phototherapy Treatments
Description: patient reported survey for Office patients only
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Office Based Phototherapy
Number analyzed (Participants) | 190
minutes
  All phototypes | 50.3 (46.7)
  Phototype I/II: number analyzed (Participants) | 79
  Phototype I/II | 53.19 (50.05)
  Phototype III/IV: number analyzed (Participants) | 93
  Phototype III/IV | 49.82 (47.43)
  Phototype V/VI: number analyzed (Participants) | 18
  Phototype V/VI | 39.72 (20.47)
Statistical Analysis 1: Comparison: Office Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Other; P-value is not applicable; Mean = 50.3, Standard Deviation 46.7
Statistical Analysis 2: Comparison: Office Based Phototherapy; Analysis for Phototypes I/II; Test type: Other; P-value is not applicable; Mean = 53.19, Standard Deviation 50.05
Statistical Analysis 3: Comparison: Office Based Phototherapy; Analysis for Phototypes III/IV; Test type: Other; P-value is not applicable; Mean = 49.82, Standard Deviation 47.43
Statistical Analysis 4: Comparison: Office Based Phototherapy; Analysis for Phototypes V/VI; Test type: Other; P-value is not applicable; Mean = 39.72, Standard Deviation 20.47

10. Secondary Outcome: DLQI (0-1)
Description: Dermatology Life Quality Index (DLQI) score of ≤1 which corresponds to no impact of dermatologic disease on quality of life. DLQI is a 10 item survey that asks patients questions about their health related quality of life on a 0-3 scale. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: The outcome measures were analyzed by skin phototype strata in addition to total subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 390 | 393
Participants
  All phototypes | 52 | 100
  Phototype I/II: number analyzed (Participants) | 169 | 181
  Phototype I/II | 25 | 56
  Phototype III/IV: number analyzed (Participants) | 180 | 170
  Phototype III/IV | 26 | 34
  Phototype V/VI: number analyzed (Participants) | 41 | 42
  Phototype V/VI | 1 | 10
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 11.97, 95% CI 2-sided [6.52 to 17.42]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 16.15, 95% CI 2-sided [7.54 to 24.75]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 5.56, 95% CI 2-sided [-2.35 to 13.46]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 21.37, 95% CI 2-sided [7.65 to 35.09]

11. Secondary Outcome: Achievement of a Minimal Clinically Important Difference (MCID) on the DLQI
Description: A difference of 4 was determined to be the MCID
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 233 | 276
Participants
  All phototypes | 130 | 188
  Phototype I/II: number analyzed (Participants) | 97 | 134
  Phototype I/II | 59 | 98
  Phototype III/IV: number analyzed (Participants) | 112 | 117
  Phototype III/IV | 56 | 74
  Phototype V/VI: number analyzed (Participants) | 24 | 25
  Phototype V/VI | 15 | 16
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.0065, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 11.68, 95% CI 2-sided [3.27 to 20.08]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.0478, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 12.31, 95% CI 2-sided [0.03 to 24.49]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.0431, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 13.25, 95% CI 2-sided [0.52 to 25.98]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.9133, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 1.50, 95% CI 2-sided [-25.50 to 28.50]

12. Secondary Outcome: Physician Global Assessment Times Body Surface Area (PGAxBSA)
Description: The difference in PGAxBSA from baseline to week 12. Values range from -500 to 500, with negative values indicating improvement in disease.
  BSA is a measure of the body surface area affected by psoriasis using the handprint method in which the palm of the entire hand approximates 1% of the body surface area. PGA is previously described. The product of the two measurements (PGA×BSA) has been investigated to assess psoriasis severity, with higher values indicating greater disease burden.
  Reference: Chiesa Fuxench et al. Validity of the simple-measure for assessing psoriasis activity (S-MAPA) for objectively evaluating disease severity in patients with plaque psoriasis. J Am Acad Dermatol 2015;73:868-7.
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 217 | 255
units on a scale
  All phototypes | -14.85 (37.75) | -23.26 (47.16)
  Phototype I/II: number analyzed (Participants) | 84 | 117
  Phototype I/II | -17.37 (33.85) | -28.04 (55.64)
  Phototype III/IV: number analyzed (Participants) | 110 | 115
  Phototype III/IV | -14.76 (38.78) | -20.06 (37.04)
  Phototype V/VI: number analyzed (Participants) | 23 | 23
  Phototype V/VI | -6.11 (45.94) | -14.94 (44.72)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.048, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = -7.90, 95% CI 2-sided [-15.73 to -0.07]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.1199, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -10.67, 95% CI 2-sided [-24.15 to 2.80]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.2953, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -5.30, 95% CI 2-sided [-15.26 to 4.66]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.5124, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -8.83, 95% CI 2-sided [-35.77 to 18.11]

13. Secondary Outcome: PGA x BSA 75%
Description: Binary outcome of achieving 75% reduction in PGA x BSA from baseline to week 12
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 217 | 255
Participants
  All phototypes | 94 | 140
  Phototype I/II: number analyzed (Participants) | 84 | 117
  Phototype I/II | 40 | 71
  Phototype III/IV: number analyzed (Participants) | 110 | 115
  Phototype III/IV | 47 | 59
  Phototype V/VI: number analyzed (Participants) | 23 | 23
  Phototype V/VI | 7 | 10
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.0173, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 10.90, 95% CI 2-sided [1.93 to 19.87]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.0662, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 13.06, 95% CI 2-sided [-0.81 to 26.94]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.1976, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 8.58, 95% CI 2-sided [-4.42 to 21.57]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.3595, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 13.04, 95% CI 2-sided [-14.60 to 40.69]

14. Secondary Outcome: PGA x BSA 90%
Description: Binary outcome of achieving 90% reduction in PGA x BSA from baseline to week 12
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 217 | 255
Participants
  All phototypes | 68 | 101
  Phototype I/II: number analyzed (Participants) | 84 | 117
  Phototype I/II | 34 | 50
  Phototype III/IV: number analyzed (Participants) | 110 | 115
  Phototype III/IV | 30 | 43
  Phototype V/VI: number analyzed (Participants) | 23 | 23
  Phototype V/VI | 4 | 8
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.0853, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 7.55, 95% CI 2-sided [-1.05 to 16.14]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.7488, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 2.26, 95% CI 2-sided [-11.54 to 16.06]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.1051, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 10.12, 95% CI 2-sided [-2.03 to 22.26]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.1792, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 17.39, 95% CI 2-sided [-7.48 to 42.27]

15. Secondary Outcome: Duration of Treatment Response During Observation Period
Description: Defined as the length of time from week 12 to the earliest of DLQI > 5 or time of initiation of a new systemic treatment or dose escalation of an existing systemic treatment, with patients who maintain DLQI <=5 5 throughout the 12 week observation period with no new systemic treatments or dose escalation censored at week 24.
Time Frame: 24 weeks after randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 96 | 177
days
  All phototypes | 74.24 (19.02) | 77.32 (16.95)
  Phototype I/II: number analyzed (Participants) | 54 | 92
  Phototype I/II | 76.37 (16.24) | 75.96 (18.16)
  Phototype III/IV: number analyzed (Participants) | 36 | 71
  Phototype III/IV | 71.17 (22.23) | 78.76 (15.39)
  Phototype V/VI: number analyzed (Participants) | 6 | 14
  Phototype V/VI | 73.5 (22.39) | 79.0 (16.64)
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p = 0.175, Regression, Linear — P-value was not adjusted for multiple comparisons; Adjusted for skin phototype; Mean Difference (Final Values) = 3.07, 95% CI 2-sided [-1.37 to 7.50]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p = 0.8904, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-6.34 to 5.51]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p = 0.0412, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 7.59, 95% CI 2-sided [0.31 to 14.88]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.5481, Regression, Linear — P-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 5.50, 95% CI 2-sided [-13.38 to 24.38]
Statistical Analysis 5: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Cox proportional hazards model for maintaining treatment response after week 12; Test type: Superiority; p = 0.458, Regression, Cox; Failure event corresponds to DLQI assessment greater than 5. Model adjusted for skin phototype; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.471 to 1.403] — Office phototherapy is the reference group

16. Secondary Outcome: Patients Receiving at Least 80% of Treatments
Description: 80% of assigned treatments is defined as 24 total treatments. Patients must have at least one treatment to be included.
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 232 | 309
Participants
  All phototypes | 62 | 202
  Phototype I/II: number analyzed (Participants) | 105 | 153
  Phototype I/II | 34 | 109
  Phototype III/IV: number analyzed (Participants) | 103 | 129
  Phototype III/IV | 22 | 82
  Phototype V/VI: number analyzed (Participants) | 24 | 27
  Phototype V/VI | 6 | 11
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis adjusted for all skin phototypes; Test type: Superiority; p < 0.0001, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 38.10, 95% CI 2-sided [30.34 to 45.86]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p < 0.0001, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 38.86, 95% CI 2-sided [27.39 to 50.33]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p < 0.0001, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 42.21, 95% CI 2-sided [30.73 to 53.68]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p = 0.2340, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 15.74, 95% CI 2-sided [-9.63 to 41.11]

17. Other Pre Specified Outcome: Safety Analysis of Skin Related Events
Description: Burns lasting 48 hours or more
Time Frame: Week 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 232 | 309
Participants
  All phototypes | 22 | 165
  Phototype I/II: number analyzed (Participants) | 105 | 153
  Phototype I/II | 11 | 77
  Phototype III/IV: number analyzed (Participants) | 103 | 129
  Phototype III/IV | 9 | 76
  Phototype V/VI: number analyzed (Participants) | 24 | 27
  Phototype V/VI | 2 | 12
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis including all skin phototypes; Test type: Superiority; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 43.96, 95% CI 2-sided [37.25 to 50.66]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Superiority; p < 0.0001, Marginal Standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 39.85, 95% CI 2-sided [30.0 to 49.70]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Superiority; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 50.18, 95% CI 2-sided [40.09 to 60.27]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Superiority; p < 0.0001, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 36.11, 95% CI 2-sided [14.35 to 57.87]

18. Other Pre Specified Outcome: Physician Global Assessment (PGA) Score of Clear/Almost Clear ("As Treated" Analysis)
Description: The outcome measure is previously described. This analysis repeats the primary outcome of PGA clear/almost clear among patients who received at least 24 treatments (i.e. 80% of assigned treatments).
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 62 | 202
Participants
  All phototypes | 32 | 95
  Phototype I/II: number analyzed (Participants) | 34 | 109
  Phototype I/II | 17 | 47
  Phototype III/IV: number analyzed (Participants) | 22 | 82
  Phototype III/IV | 14 | 42
  Phototype V/VI: number analyzed (Participants) | 6 | 11
  Phototype V/VI | 1 | 6
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis including all skin phototypes; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.1773, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -5.2, 95% CI 2-sided [-19.4 to 9.0]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.4073, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -6.88, 95% CI 2-sided [-26.09 to 12.33]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.8247, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -12.42, 95% CI 2-sided [-35.24 to 10.41]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.0133, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 37.88, 95% CI 2-sided [-4.01 to 79.77]

19. Other Pre Specified Outcome: Impact of Dermatological Disease on Quality of Life ("As Treated" Analysis)
Description: The outcome measure is previously described. This analysis repeats the primary outcome of DLQI <=5 among patients who received at least 24 treatments (i.e. 80% of assigned treatments).
Time Frame: 12 weeks after randomization or earlier at discontinuation of phototherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 62 | 202
Participants
  All phototypes | 39 | 140
  Phototype I/II: number analyzed (Participants) | 34 | 109
  Phototype I/II | 22 | 79
  Phototype III/IV: number analyzed (Participants) | 22 | 82
  Phototype III/IV | 14 | 53
  Phototype V/VI: number analyzed (Participants) | 6 | 11
  Phototype V/VI | 3 | 8
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Overall analysis including all skin phototypes; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.002, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 6.52, 95% CI 2-sided [-7.11 to 20.14]
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes I/II; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.0137, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 7.77, 95% CI 2-sided [-10.35 to 25.89]
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes III/IV; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.1656, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 1.0, 95% CI 2-sided [-21.61 to 23.61]
Statistical Analysis 4: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Analysis for Phototypes V/VI; Test type: Non-Inferiority — Statistical inference was based on non-inferiority principles using a non-inferiority margin of 15%; p = 0.1225, Marginal standardization — P-value was not adjusted for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = 22.73, 95% CI 2-sided [-25.16 to 70.62]

20. Other Pre Specified Outcome: Dichotomized DLQI Beyond Week 12
Description: Number of participants that had a DLQI <= 5 at week 16, week 20, and week 24
Time Frame: From Week 12 to Week 24
Population: The number analyzed per time point differ due to missing DLQI response
Measure: Count of Participants; unit: Participants
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
Number analyzed (Participants) | 169 | 233
Participants
  Week 16 | 90 | 150
  Week 20: number analyzed (Participants) | 161 | 188
  Week 20 | 88 | 118
  Week 24: number analyzed (Participants) | 160 | 215
  Week 24 | 105 | 139
Statistical Analysis 1: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Difference of proportion at week 16. Calculated using contrasts of predictive margins following logistic regression with robust variance estimators via generalized estimating equations and exchangeable correlation. Missing data for DLQI are imputed using multiple imputation via chained equations (10 imputations), and the estimates are combined using standard rules; Test type: Superiority; p = 0.0183, Marginal contrast; Risk Difference (RD) = 0.105, 95% CI 2-sided [0.018 to 0.192] — Positive values indicate higher proportion in the home group
Statistical Analysis 2: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Difference of proportion at week 20. Calculated using contrasts of predictive margins following logistic regression with robust variance estimators via generalized estimating equations and exchangeable correlation. Missing data for DLQI are imputed using multiple imputation via chained equations (10 imputations), and the estimates are combined using standard rules; Test type: Superiority; p = 0.177, Marginal contrast; Risk Difference (RD) = 0.064, 95% CI 2-sided [-0.029 to 0.158] — Positive values indicate higher proportion in the home group
Statistical Analysis 3: Comparison: Office Based Phototherapy vs Home Based Phototherapy; Difference of proportion at week 24. Calculated using contrasts of predictive margins following logistic regression with robust variance estimators via generalized estimating equations and exchangeable correlation. Missing data for DLQI are imputed using multiple imputation via chained equations (10 imputations), and the estimates are combined using standard rules; Test type: Superiority; p = 0.815, Marginal contrast; Risk Difference (RD) = -0.011, 95% CI 2-sided [-0.101 to 0.079] — Positive values indicate higher proportion in the home group

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for up to 24 weeks from beginning of study.
Arm/Group | Office Based Phototherapy | Home Based Phototherapy
All-Cause Mortality (participants affected / at risk) | 0/390 | 1/393
Serious Adverse Events (participants affected / at risk) | 4/390 | 3/393
Other Adverse Events (participants affected / at risk) | 22/390 | 165/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Office Based Phototherapy (N=390) | Home Based Phototherapy (N=393)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hospitalization for infected wounds (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization for substance abuse treatment (General disorders) | 0 (0) | 1 (1)
Severe neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization for blood pressure (General disorders) | 0 (0) | 1 (1)
Seen in ER for chest pain (General disorders) | 1 (1) | 0 (0)
Death (Covid-19 related) (Infections and infestations) | 0 (0) | 1 (1)
Malnutrition resulting in hospitalization (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Office Based Phototherapy (N=390) | Home Based Phototherapy (N=393)
Burns from phototherapy treatment (Skin and subcutaneous tissue disorders) | 22 (46) | 165 (466) — Treatments that caused erythema > 48 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT03726489/Prot_SAP_000.pdf